CLINICAL TRIAL: NCT05070442
Title: Diet Improvement Through Normative Experimentation
Acronym: DINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NIHA-2018-002 (Study 2)
Record Dates: First submitted 2021-09-20; First posted 2021-10-07 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Diet Quality
Keywords: Nutri-Score labels; Social norms; Peer comparison; Financial incentives; Loss aversion; Online grocery shopping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Arm 1) (No Intervention): Participants will experience an unmodified version of NUSMart which replicates the traditional shopping experience of online grocery stores.
- Norms Arm (Arm 2) (Experimental): Participants will experience a modified version of NUSMart with norm-based messaging and peer comparison features enabled. Nutri-Score labels will be enabled and displayed on all products within the store. A floating side panel will provide a visual indicator of the participants' average weighted Nutri-Score.
  Interventions: Behavioral: Norm-based messaging and peer comparison features
- Norms and Incentive Arm (Arm 3) (Experimental): Same as Arm 2, except participants are notified that they have been awarded an additional $5 towards their participation reimbursement. However, this additional $5 will be forfeited if their basket average weighted Nutri-Score falls below the average of their peers'. (Financial incentive leveraging on loss aversion).
  Interventions: Behavioral: Norm-based messaging and peer comparison features; Behavioral: Financial Incentives leveraging on loss aversion

INTERVENTIONS:
Behavioral: Norm-based messaging and peer comparison features — Participants are shown a version of NUSMart which includes Nutri-Score labels that are enabled and displayed besides all the products in the store. Additionally, they are shown a video that gives them background information about Nutri-Score labels and describes the following features enabled in this intervention:
  * Norm-based messaging will be displayed in the form of a happy or sad emoticon based on whether the participant's current basket average Nutri-Score (weighted by number of servings) is above or below "other shoppers" (Nutri-Score=3.98).
  * Peer comparison will be implemented as a vertical ruler display of the participant's current basket average Nutri-Score (weighted by number of servings) as well as that of their "peers".
  Nutri-Score=3.98 was chosen as it is 10% better than the mean Nutri-Score of baskets purchased by participants in the Nutri-Score labelled intervention arm of a prior study.
  Arms: Norms Arm (Arm 2); Norms and Incentive Arm (Arm 3)
Behavioral: Financial Incentives leveraging on loss aversion — Participants are informed that they have received an additional $5 towards their participant reimbursement. However, this amount will be forfeited if they check-out with a basket average Nutri-Score (weighted by the number of servings) that falls below the average Nutri-Score of "other shoppers" i.e. 3.98. An indicator on the screen that informs the participants of this potential forfeiting will be included.
  Arms: Norms and Incentive Arm (Arm 3)

SUMMARY:
This study aims to use a three-arm randomized control trial (RCT) implemented in a fully functional experimental online grocery store, to explore the effects of two low-cost information and incentive-based strategies. These strategies comprise of injunctive norm-based messaging and the use of financial incentive leveraging on loss aversion to encourage the purchase of healthy foods. The investigators have set up a store wherein products may be purchased by participants and subsequently delivered to homes in some of the conditions. This increases the external validity of these interventions and enables investigators to establish greater confidence in their generalizability.

DETAILED DESCRIPTION:
The Asia-Pacific is faced with an epidemic of rising rates of chronic disease. Poor diet quality is a demonstrated risk factor for non-communicable diseases. Excess intake of calories, saturated fat and sodium increases the risk of obesity, heart disease, diabetes, and other chronic conditions.

Behavioral economics has emerged as a promising strategy to increase the effectiveness of interventions aimed to address risk factors for non-communicable diseases (NCDs). Yet, there is a gap in knowledge concerning how norm-based messaging and peer influence interventions can be implemented to improve diet quality.

Using a three-arm randomized trial with a 3x3 crossover design, investigators aim to determine whether norm-based messaging and peer comparisons, with or without financial incentives, improve diet quality.

Each participant will be exposed to all of the following intervention arms in random order:

Arm 1: Control arm. Participants will experience an unmodified version of NUSMart which replicates the traditional shopping experience of online grocery stores.

Arm 2: Participants will experience a modified version of NUSMart with norm-based messaging and peer comparison features enabled. Nutri-Score labels will be enabled and displayed on all products within the store. A floating side panel will provide a visual indicator of the participants' average weighted Nutri-Score.

Arm 3: Same as Arm 2, except participants are notified of an additional $5 reward towards participation reimbursement. However, this additional $5 will be forfeited if the basket average weighted Nutri-Score falls below the average of participants' peers'. (Financial incentive leveraging on loss aversion).

Investigators hypothesize the following:

Primary hypothesis: Diet quality, as measured by mean Nutri-Score weighted by number of servings of all basket items, will be greatest when exposed to the intervention with norm-based messaging with incentive (Arm 3), followed by the intervention with norm-based messaging without the incentive (Arm 2), followed by Control (Arm 1).

Investigators will test this hypothesis in total, and separately for foods and beverages given Singapore's focus on reducing intake of sugar-sweetened beverages.

ELIGIBILITY:
Inclusion Criteria:

* Singapore resident
* Age 21 and above
* Must be the primary weekly grocery shopper in their household

Exclusion Criteria:

* Non-Singapore resident
* Non-primary grocery shopper in their household
* Less than 21 years old

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Diet Quality | After completion of data collection, an average of about 5 months
  Diet quality, as measured by raw Nutri-Score points (-15 to 40) weighted by number of servings of all basket items. Here, a smaller value means a better outcome. Raw Nutri-Score is measured according to the guidelines from the Sante Publique France.

SECONDARY OUTCOMES:
Average Nutri-Score | After completion of data collection, an average of about 5 months
  Average Nutri-Score (1 to 5) weighted by number of servings of all basket items. Here, a higher value means a better outcome. This is calculated by converting Nutri-Score letters to numbers such that Nutri-Score E is 1, D is 2 and so on till Nutri-Score A which is 5.
Average Calories | After completion of data collection, an average of about 5 months
  Average calories per shopping trip.
Average Sodium | After completion of data collection, an average of about 5 months
  Average sodium per shopping trip.
Average Sugar | After completion of data collection, an average of about 5 months
  Average sugar per shopping trip.
Average Fat | After completion of data collection, an average of about 5 months
  Average fat per shopping trip.
Average Saturated Fat | After completion of data collection, an average of about 5 months
  Average saturated fat per shopping trip.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, PhD MHA, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No